CLINICAL TRIAL: NCT00720707
Title: Coronally Advanced Flap in Combination With Acellular Dermal Matrix With or Without Enamel Matrix Derivatives for Root Coverage
Brief Title: Coronally Advanced Flap in Combination With Acellular Dermal Matrix and Enamel Matrix Derivatives for Root Coverage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tabriz University (Other)
Responsible Party: Dr. Reza Pourabbas, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 841
Record Dates: First submitted 2008-07-22; First posted 2008-07-23 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-07

CONDITIONS: Gingival Recession
Keywords: Coronally advanced flap; gingival recession; enamel matrix protein; acellular dermal matrix; root coverage
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm; enamel matrix proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (CAF+ADM+EMD) (Experimental): using coronally advanced flap (CAF) in combination with acellular dermal matrix (ADM) with enamel matrix derivatives (EMD).
  Interventions: Procedure: CAF+ADM+EMD
- (CAF + ADM) (Active Comparator): root coverage procedure by using a coronally advanced flap (CAF) in combination with acellular dermal matrix (ADM)
  Interventions: Procedure: CAF+ADM

INTERVENTIONS:
Procedure: CAF+ADM+EMD — using coronally advanced flap (CAF) in combination with acellular dermal matrix (ADM) with enamel matrix derivatives (EMD).
  Other Names: Alloderm®; Emdogain®
  Arms: (CAF+ADM+EMD)
Procedure: CAF+ADM — using coronally advanced flap (CAF) in combination with acellular dermal matrix (ADM) without enamel matrix derivatives (EMD) for root coverage procedures.
  Other Names: Alloderm®; Emdogain®
  Arms: (CAF + ADM)

SUMMARY:
The aim of this study is to compare the clinical outcomes of root coverage procedures, using coronally advanced flap in combination with acellular dermal matrix with or without enamel matrix derivatives .

DETAILED DESCRIPTION:
coverage of gingival recession defects has been considered as a matter of interest for dental practitioners.subjects with a paired gingival recession defect will be selected from the patients who sought dental treatment at our department.Random allocation of the treatment sites to test (CAF+ EMD+ADM) and control (CAF + ADM) groups will be performed by a person who is external to the study and using a computerized selection of random numbers for allocation of the study groups.The parameters of the study are as following items: probing depth( PD), clinical attachment level (CAL), width of keratinized tissue (WKT), recession depth from cemento- enamel junction (RD), recession width (RW), distance between mucogingival junction and the stent (MGJ), Plaque (PI) and gingival (GI) indices and root coverage percentage (RC) and the patients will be followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Having no systemic disease affecting the periodontium,
* No contraindication for elective surgery,
* Adequate oral hygiene ,
* No previous surgical attempts for root coverage at the studying sites,
* Vital teeth and signing a witness letter.

Exclusion Criteria:

* Smoking, presence of a restorations on tooth surface for test and control teeth,
* Pregnancy,
* Being under treatment with steroids,
* Peri-apical infection,
* Indication for antibiotic prophylaxis prior to dental treatments

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
the percentage of root coverage | at baseline, 2 and 6 months after treatment.

SECONDARY OUTCOMES:
clinical attachment level, width of keratinized gingiva ant the position of mucco-gingival junction following root coverage procedures | 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Reza Pourabbas, DDS, Principal Investigator — Tabriz University (Medical Sciences)
Locations (1):
- Faculty of Dentistry- Tabriz University of Medical Sciences, Tabriz, East Azerbaijan Province, Iran